CLINICAL TRIAL: NCT03913078
Title: Comparative Effectiveness of Social Physical Play and Traditional Exercise Programming
Acronym: PlayFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Professor of Medicine and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HL142679; R33HL142679 (NIH)
Record Dates: First submitted 2019-04-09; First posted 2019-04-12 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Group Fitness (Traditional); Group Fitness (Game Play-based)
Keywords: fitness; exercise; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Increases in perceived enjoyment lead to increases in physical activity adherence which lead to increases in physical fitness
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants are aware of the two different exercise conditions and accept randomization into either of the two. The investigator and outcomes assessor are masked, but participant is aware of group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Fitness (Active Comparator): Subjects will be offered several sessions per week of a traditional group fitness program led by a trained group leader.
  Interventions: Behavioral: Group Fitness
- PlayFit (Active Comparator): Subjects will be offered several sessions per week of a modified sports fitness program, led by a trained group leader.
  Interventions: Behavioral: PlayFit

INTERVENTIONS:
Behavioral: Group Fitness — Traditional Group Fitness consisting of aerobic and strength exercises performed in a group setting and led by a trained instructor.
  Arms: Group Fitness
Behavioral: PlayFit — Modified sports fitness exercise program consisting of games played in groups and led by a trained instructor.
  Arms: PlayFit

SUMMARY:
This study will compare the impact of traditional group fitness versus a game-based fitness program, designed to maximize enjoyment, on physical fitness.

DETAILED DESCRIPTION:
Fewer than 1 in 10 middle-aged US adults get the recommended amount of aerobic physical activity (PA), greatly increasing their chances of heart disease and stroke. There are over 50 million adults with fitness center memberships, which are used only once per month and, after joining new programs, people quickly stop coming. While many barriers to PA have been cited (e.g., time, cost), the investigators believe that a key, modifiable, and underappreciated barrier is that most adults simply do not enjoy physical activity enough to do it regularly. Studies consistently observe that people who enjoy physical activity more are more likely to be more active in the future. Despite this consistent observation, the investigators are not aware of studies that ask "Would an adult PA program designed to maximize enjoyment increase PA adherence and fitness?". In 2015, our team set out to design an exercise program for adults that maximized enjoyment. Taking inspiration from Pickleball, a popular game of modified tennis, our team created PlayFit. PlayFit is an exercise program in which adults come together three times each week to play a range of sports, all modified to 1) reduce effort (e.g., smaller playing area), 2) reduce injuries (e.g., lightweight low-pressure balls) and 3) reduce competitiveness (e.g., teams chosen randomly, minimize physical contact, no keeping score). Pilot work in the summer of 2016 with 22 adults identified five modified sports that all had Metabolic Equivalent (MET) levels between 5.5 and 6.5 and high satisfaction scores (average of 8.0 out of 10). More importantly, the comments suggest that the investigators have created a social, enjoyable experience: "that was SO much fun", "I've never had so much fun playing soccer". People liked "the laughter during the games", "no pressure, not competitive" and that "it's not about ability, it's just about having fun with people".

In this study, the investigators initially proposed testing whether PlayFit would lead to greater fitness gains, compared to group fitness, to help providers understand in a way that helps providers and fitness center staff understand: "What exercise program should I recommend to promote long-term adherence and fitness?". All subjects were to be expected to exercise three-times weekly for 60 minutes for 12 months. The investigators planned to randomly assign 360 adults to two conditions: 1) Group Fitness activities and 2) PlayFit. The investigators hypothesized that both PlayFit and Group Fitness would increase Maximum Oxygen Uptake (V02max) significantly at 6 months but, after 12 months, mediated by greater enjoyment and higher adherence, participants randomized to PlayFit would have greater fitness and activity gains at 12 months than Group Fitness. The results of this study would have the potential to help patients, providers and fitness center directors by answering the question: "What exercise program should be recommended to sedentary adults in order to promote long-term adherence and fitness?"

Although we originally intended for data collection to conclude by 2021, human-subjects research was largely prohibited throughout 2020 due to the SARS-CoV-2 pandemic. Near the end of 2020 we began to conduct outdoor-only activities. Indoor human-subjects research continued to be restricted throughout 2020 and early 2021.

Once large-scale research restrictions were lifted, recruitment and baseline testing resumed in May 2021, with the first new cohorts beginning in their respective sessions in August 2021. Unfortunately, all human-subjects research was again prohibited for approximately 45 days during January and February 2022. For several reasons, including the likely deconditioning of participants during the pause, that several participants responded that they were unwilling or fearful to return given the perceived health risks, and that some community partners were no longer willing to host the PA sessions during the pandemic, we concluded that our best course of action was to analyze data up to the most recent measurement timepoint preceding this 45-day mandated pause in data collection (month 3).

This decision meant that we were unable to test our original hypotheses. For example, only baseline cardiorespiratory fitness and accelerometry data were available, as the second time point to collect these data was to occur at month 6. However, analyses for group session adherence were possible, as these data were collected continuously throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Sedentary (<90 minutes of self-reported moderate-vigorous activity each week)
* Health care provider must give permission.

Exclusion Criteria:

* History of heart disease, stroke or chest pain.
* Participating in another research study involving physical activity or weight loss.
* Planning to have surgery or move in the next year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sciamanna, MD, MPH, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Final, clean, data filed will be uploaded to a publicly available site (e.g., ISPSR), within 12 months of finishing study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 12 months of completing the final follow-up visit on the last study subject.
URL: https://www.icpsr.umich.edu/icpsrweb/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 26 participants consented to participate in the study, but did not complete baseline measures, and were therefore not allocated to a study arm.
Period: Overall Study
Arm/Group | Group Fitness | PlayFit
Started | 200 | 205
Completed | 200 | 205
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Fitness | PlayFit | Total
Number analyzed (Participants) | 200 | 205 | 405
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (7.2) | 39.7 (7.6) | 39.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 146 | 292
  Male | 54 | 59 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 10 | 23
  Not Hispanic or Latino | 174 | 182 | 356
  Unknown or Not Reported | 13 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 11 | 20 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 12 | 31
  White | 144 | 146 | 290
  More than one race | 7 | 9 | 16
  Unknown or Not Reported | 17 | 17 | 34
Region of Enrollment [Number; unit: participants]
  United States | 200 | 205 | 405
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: All participants contributing data were included in this analysis.
  kg/m^2
    number analyzed (Participants) | 186 | 181 | 367
    (all) | 33.0 (10.1) | 33.1 (10.0) | 33.0 (10.0)
VO2 Maximum [Mean (Standard Deviation); unit: ml/kg/min] — Population: As indoor activities were restricted by the SARS-CoV-2 pandemic, some participants were unable to complete VO2 maximum testing.
  ml/kg/min
    number analyzed (Participants) | 49 | 92 | 141
    (all) | 23.7 (5.1) | 25.1 (9.0) | 24.4 (7.4)
MVPA [Mean (Standard Deviation); unit: minutes per week] — Moderate-to-vigorous physical activity, measured via accelerometry in minutes per week Population: The ability to distribute accelerometers was limited by the SARS-CoV-2 pandemic.
  minutes per week
    number analyzed (Participants) | 82 | 84 | 166
    (all) | 164.1 (92.0) | 168.1 (88.0) | 166.1 (89.7)

OUTCOME MEASURES:

1. Primary Outcome: Session Attendance
Description: Adherence to the intervention sessions was collected by the PlayFit and Group Fitness group leaders during each session using a REDCap attendance survey.
Time Frame: Duration of participation in study, up to 1 year
Population: All participants that were assigned to an arm are included in this analysis, even if they never attended a session
Measure: Mean (Standard Deviation); unit: Percentage of possible sessions attended
Arm/Group | Group Fitness | PlayFit
Number analyzed (Participants) | 200 | 205
Percentage of possible sessions attended | 12.3 (15.5) | 10.4 (13.0)

2. Post Hoc Outcome: Total Possible Sessions
Description: This is the total number of sessions that each participant was potentially able to attend.
Time Frame: Duration of participation in study, up to 1 year
Measure: Mean (Standard Deviation); unit: Possible sessions
Arm/Group | Group Fitness | PlayFit
Number analyzed (Participants) | 200 | 205
Possible sessions | 104.3 (49.7) | 110.0 (55.9)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected monthly for the duration of participation in the study, up to 1 year. This time period varied by participant due to the impact of the SARS-CoV-2 pandemic.
Description: Injuries and other adverse events were assessed monthly using a self-report questionnaire that consisted of 7-items focusing on injury location and severity.
Arm/Group | Group Fitness | PlayFit
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/205
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/205
Other Adverse Events (participants affected / at risk) | 19/200 | 38/205
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Fitness (N=200) | PlayFit (N=205)
Musculoskeletal Injury (Musculoskeletal and connective tissue disorders) | 18 (23) | 37 (50)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Human-subjects research was largely prohibited throughout 2020 and early 2021 due to the SARS-CoV-2 pandemic. Large-scale research restrictions were lifted in May 2021. All human-subjects research was again prohibited during January and February 2022. After that pause, participants were unwilling to return given the perceived health risks and community partners were no longer willing to host the PA sessions during the pandemic. Full participation in the trial as planned was then not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT03913078/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03913078/ICF_001.pdf